CLINICAL TRIAL: NCT01091610
Title: Work Related Injuries Among Prehospital Emergency Medical Staff, a Retrospective, Observational Study
Brief Title: Work Related Injuries Among Prehospital Emergency Medical Staff, an Observational Study
Status: Withdrawn | Type: Observational
Why Stopped: no collaboration
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Sammelstelle der Statistik der Unfallversicherungen (SSUV), Luzern (Unknown)
Responsible Party: Dr. med. Kay Stricker, Universitätsklinik für Anästhesiologie und Schmerztherapie, Inselspital, Bern University Hospital and University of Bern, CH 3010 Bern
Other Study IDs: KEK21-01-10
Record Dates: First submitted 2010-03-21; First posted 2010-03-24 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2011-03

CONDITIONS: Wounds and Injuries; Accidents, Occupational
Keywords: retrospective study; wounds and injuries/epidemiology; emergency medical technicians; human; emergency medical services; ambulance; health personnel; emergency medicine; risk factors
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: all emergency medical staff having suffered an accident during work
  Interventions: Other: no intervention
- 2: non emergency medical personnel having suffered an injury due to a medical mission, e.g. transported patient having suffered additional injury due to an ambulance accident or collision of an ambulance with another vehicle.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — purely observational retrospective study. no interventions are planned.

SUMMARY:
Ambulance personnel often work in a dangerous environment and work related injuries of emergency medical staff have repeatedly been documented. However, only case reports are published and no data exist about the incidence and type of work related injuries of ambulance personnel.

Aims:

The primary aim of the study is to assess the incidence (number of new injuries per 100'000 emergency missions or per 1'000 flying hours) and type of work related injuries among prehospital emergency personal. The secondary aims are to identify risk factors associated with work related injuries and to compare the risk of injury to other groups of professionals such as hospital nurses, policemen or fire-fighters.

DETAILED DESCRIPTION:
Background

Background:

Staff of emergency medical missions is at high risk of work-related injuries. Over 8 % of emergency medical staff have been reported to be victims of work-related injuries, leading to a time away from work of 9.4 %. Others have reported a rate of 5 - 25 accidents per 100'000 flight hours or 55 per 100'000 road ambulance transports. A ten year retrospective analysis of US public roadways identified 331 accidents with 405 fatalities and 838 injuries. Speed of work, unknown work surroundings, difficult working conditions such as poor lighting and tight work environment may all contribute to injuries. While mishaps and unintentional injuries cause most incidents, frank assaults pose additional threats to medical staff. In the US the injury rate for EMS workers are higher than rates reported by the department of labour for any other industry. Most commonly reported injuries include strains and sprains, however, permanent disabilities and fatal injuries have been reported. Even though the medical profession's first duty is to do no harm, innocent bystanders have repeatedly been victims of ambulance crashes. In fact, one study reported a greater burden of injury on persons not in the ambulance. While emergency medical work pose some intrinsic risks to patients and workers, several risk factors have been identified which are associated with increased risk of incapacitating or fatal injuries, e.g., positioning in the rear of an ambulance or improper restrains, younger EMS professionals and sleeping problems and while on non-emergency travels. Inadequate restrains pose a particular risk in paediatric emergency transport.

No data for work-related injuries have been reported for prehospital medical crew in Europe.

Aims:

The primary aim of the study is to assess the incidence (number of new injuries per 100'000 emergency missions or per 1'000 flying hours) and type of work related injuries among prehospital emergency personal. The secondary aims are to identify risk factors associated with work related injuries and to compare the risk of injury to other groups of professionals such as hospital nurses, policemen or fire-fighters.

Setting:

Prehospital emergency medical services (EMS) in Switzerland, including ground, air and water-related ambulance services. All certified ambulance services for air, traffic and water accidents are eligible for participation and will be contacted and invited to participate. Additional supporting rescue companies such as rescue squad of the Swiss Alpine Club or of a ski resort as well as lay rescuers will not be included in the analysis. All accidents on medical missions of a prolonged period are analysed. Depending on the available data in the different ambulance services, the study period may extend from at least one year up to a maximum of 10 years.

Methods:

Incidents are defined as:

* an unintentional (i.e. accident) or intentional (i.e. assault) injury during an emergency medical mission leading to leave from work, including:

  * EMS personal,
  * innocent bystanders or
  * additional injuries to patients transported;
* a needle stick injury, even if it will not lead to a leave from work;
* a leave from work due to a severe psychological distress during an emergency mission, e.g. death of a child

Medical reasons (e.g. common flu, chronic back pain) resulting in leave from work are not considered as incidents and will not be included.

Severity of injury will be stratified according to the KABCO classification as suggested previously (K: killed, A: incapacitating injury, B: non-incapacitating injury, C: possible injury, O: no apparent injury).

Incidents will be analysed according to parameters related to an ambulance organisation, type of emergency mission and injuries to patients, EMS personal and innocent bystanders. Since the prevalence of accidents or near misses is expected to be low, a large number of emergency missions of a large time span must be investigated. To allow a timely analysis, data will be gathered retrospectively. The data of the victims (cases, i.e. ambulance worker) will be collected anonymously. Cases will be identified using the accident number (Schadennummer) and the UVG (Unfallversicherungsgesetz) insurer. Personal data will thus be anonymous at the study centre in Bern.

Data evaluation and statistics:

In a first step the total incidence of work-related injuries (number of new injuries divided by number of missions or divided by number of flying hours) will be determined as primary endpoint among street, air and sea ambulance services in Switzerland. Descriptive statistics will be used.

Risk factors, i.e. secondary endpoints, will be analyzed using univariable and multivariable multilevel linear regression models with three levels: 1. ambulance organization, 2. ambulance mission and 3. victim. Possible risk factors may include for:

* ambulance organization:

  * type of ambulance organization, (ground, air, sea)
  * geographical region of the ambulance organization (German, French, Italian-romansch speaking region of Switzerland)
  * rural - urban setting
  * hospital association of ambulance service
  * number of collaborators at ambulance service
  * number of missions per year
* mission:

  * time of day
  * weekday
  * time of year
  * weather conditions
  * duration of mission
  * type of accident (unintentional accident, assault, psychological "injury")
  * phase of mission (during approach, on site of accident, on way to hospital, during hand-over / on hospital ground, on way home)
  * type of mission (primary mission, i.e. direct approach to accident, secondary mission (interhospital transfer).
  * with / without special signal, i.e. signal and lights
* Victim associated:

  * Age at the time of accident
  * gender
  * years of on the job experience
  * role during the accident-related rescue mission (driver, paramedic, pilot,…), position at time of accident (driver compartment, patient compartment,…)
  * part-time, fulltime employment
  * number of mission per collaborator and per year
  * patient characteristics (patient to be transported suffered additional injury, patient escort e.g. parent of child-patient, member of rescue team, bystander)
  * degree of injury (deceased, permanent injury, non-permanent injury, possible injury, uninjured)
  * duration of leave from work
  * position at the time of accident (driver compartment, patient compartment, outside vehicle, in / on other vehicle)
  * innocent bystander
  * patient to be transported

In a second step the comparison with other professional groups, e.g. hospital nurses, policemen or fire-fighters will be performed. The data of the first step will allow to perform a sample size calculation for future research.

Objective

Aims:

The primary aim of the study is to assess the incidence (number of new injuries per 100'000 emergency missions or per 1'000 flying hours) and type of work related injuries among prehospital emergency personal. The secondary aims are to identify risk factors associated with work related injuries and to compare the risk of injury to other groups of professionals such as hospital nurses, policemen or fire-fighters.

Methods

Prehospital emergency medical services (EMS) in Switzerland. All certified ambulance services for air, traffic and water accidents are eligible for participation and will be contacted and invited to participate. All accidents on medical missions of a prolonged period are analysed.

Incidents are defined as:

* an unintentional (i.e. accident) or intentional (i.e. assault) injury during an emergency medical mission leading to leave from work, including:

  * EMS personal,
  * innocent bystanders or
  * additional injuries to patients transported;
* a needle stick injury, even if it will not lead to a leave from work;
* a leave from work due to a severe psychological distress during an emergency mission

ELIGIBILITY:
Inclusion Criteria:

* human
* leave from work
* work related mortality
* work related injury
* needle stick injury
* psychological distress
* innocent bystander
* unintentional injury
* intentional injury
* emergency mission

Exclusion Criteria

* medical reason
* chronic illness
* non-work related injury
* non-work related mortality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all ambulance companies in Switzerland (including air, ground and water associated) will be contacted to provide data of their personnel of the past 10 years. All accidents leading to leave from work will be analyzed according to parameters concerning the ambulance organisation, the person and the emergency mission. In addition, data of additionally injured non-medical persons due to an emergency mission will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05

PRIMARY OUTCOMES:
overall incidence of injuries and mortality | 10 years

SECONDARY OUTCOMES:
risk factors for injuries | 10 years
incidence of additional injuries to others | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kay H Stricker, MD, Study Chair — Department of anaesthesiology and pain medicine, Bern University Hospital; Martin Luginbühl, MD, Study Director — Department of anaesthesiology and pain medicine, Bern University Hospital
Locations (2):
- Switzerland (2):
  - department of anaesthesiology and pain medicine, Bern University Hospital, Bern,, Bern, Canton of Bern
  - SSUV Sammelstelle für die Statistik der Unfallversicherungen, Lucerne, Canton of Lucerne

REFERENCES:
- [Background] Maguire BJ, Hunting KL, Smith GS, Levick NR. Occupational fatalities in emergency medical services: a hidden crisis. Ann Emerg Med. 2002 Dec;40(6):625-32. doi: 10.1067/mem.2002.128681. PMID 12447340
- [Background] Maguire BJ, Hunting KL, Guidotti TL, Smith GS. Occupational injuries among emergency medical services personnel. Prehosp Emerg Care. 2005 Oct-Dec;9(4):405-11. doi: 10.1080/10903120500255065. PMID 16263673
- [Background] Studnek JR, Ferketich A, Crawford JM. On the job illness and injury resulting in lost work time among a national cohort of emergency medical services professionals. Am J Ind Med. 2007 Dec;50(12):921-31. doi: 10.1002/ajim.20516. PMID 17918231
- [Background] Flabouris A, Runciman WB, Levings B. Incidents during out-of-hospital patient transportation. Anaesth Intensive Care. 2006 Apr;34(2):228-36. doi: 10.1177/0310057X0603400216. PMID 16617646
- [Background] Kahn CA, Pirrallo RG, Kuhn EM. Characteristics of fatal ambulance crashes in the United States: an 11-year retrospective analysis. Prehosp Emerg Care. 2001 Jul-Sep;5(3):261-9. doi: 10.1080/10903120190939751. PMID 11446540
- [Background] Greene J. Rising helicopter crash deaths spur debate over proper use of air transport. Ann Emerg Med. 2009 Mar;53(3):15A-17A. doi: 10.1016/j.annemergmed.2009.01.007. No abstract available. PMID 19244622
- [Background] Johnson TD, Lindholm D, Dowd MD. Child and provider restraints in ambulances: knowledge, opinions, and behaviors of emergency medical services providers. Acad Emerg Med. 2006 Aug;13(8):886-92. doi: 10.1197/j.aem.2006.03.562. Epub 2006 Jul 6. PMID 16825667
- [Background] Becker LR, Zaloshnja E, Levick N, Li G, Miller TR. Relative risk of injury and death in ambulances and other emergency vehicles. Accid Anal Prev. 2003 Nov;35(6):941-8. doi: 10.1016/s0001-4575(02)00102-1. PMID 12971929